CLINICAL TRIAL: NCT04750356
Title: SARS-CoV-2 Longitudinal Study: Understanding Susceptibility, Transmission and Disease Severity
Brief Title: SARS-CoV-2 (COVID-19) Longitudinal Study: Understanding Susceptibility, Transmission and Disease Severity (Legacy Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Francis Crick Institute (Other)
Responsible Party: Sponsor
Other Study IDs: UCLH 134617
Record Dates: First submitted 2021-01-28; First posted 2021-02-11 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: SARS-CoV Infection
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blod samples and nasal and throat swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort A1: Healthcare workers and patients that have previously undertaken a swab or serology test to detect for the presence of SARS-CoV-2. Without the need to seek retrospective consent for the SARS CoV 2 Longitudinal Study, residual samples and derivatives from the Crick COVID -9 Consortium Testing centre and data will be used for the study
- Cohort A2: 3,000 SARS-CoV-2 positive and 3,000 SARS-CoV-2 negative participants (randomly selected) from cohort A1 will be prospectively consented to the study. In addition, vaccine status will also be used to stratify the participants and recruit to the study.
- Cohort B: Employees at participating centres including but not limited to UCLH and The Francis Crick Institute who have their serology tested and/or are swabbed for viral (SARS-CoV-2 and seasonal viruses) detection as well as participants who are vaccinated will be prospectively consented to the study.
- Cohort C: Individuals recruited to other REC approved research studies where their samples are processed by the Crick COVID 19 Consortium Testing centre will also be consented in their existing study to allow the use of leftover study samples already collected and to be collected, for use in this longitudinal study.

SUMMARY:
The study aims to investigate SARS-CoV-2 susceptibility, transmission and disease severity in healthcare workers and patients.

Residual specimens from an existing collection of samples in viral inactivating buffer and derivatives and serum from the Crick COVID-19 Consortium Testing centre (Cohort A1) and additional biological material collected prospectively (Cohorts A2 and B) will be used for research into SARS-CoV-2 transmission, evolution and immune control. This testing centre is a partnership between UCLH and The Francis Crick Institute to provide COVID 19 RT PCR testing for healthcare workers (HCWs) and patients in London Hospitals and care homes. A third group (Cohort C) of the study will allow for collaborative work with other REC approved research studies that have used the Crick COVID-19 Consortium Testing centre and will involve the use of study samples already collected from each study to be analysed under the SARS-CoV-2 Longitudinal Study end points

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have previously provided nasal throat swab samples for SARS-CoV-2 testing at the Crick COVID 19 Consortium Testing centre.
* ≥18 years of age
* To enrol in the SARS-CoV-2 positive cohort of the study, the participant should have a positive RT qPCR result
* Employees based at the participating sites including who had their serology and/or swab tested (for recruitment to Cohort B)
* Participants enrolled in other studies who had their samples processed by using the Crick COVID 19 Consortium Testing centre (for recruitment to Cohort C).
* Written informed consent (except Cohort A1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who have previously provided samples for SARS-CoV-2 testing at the Crick COVID 19 Consortium Testing centre
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 susceptibility in healthcare workers and patients | 24 months
  To investigate SARS-CoV-2 susceptibility by examining the number of positive SARS-CoV-2 result per participant
SARS-CoV-2 transmission in healthcare workers and patients | 24 months
  To investigate SARS-CoV-2 transmission by analysis of samples sequencing data from each study centre and across study centres
SARS-CoV-2 severity in healthcare workers and patients | 24 months
  To investigate SARS-CoV-2 severity by review of symptom severity
SARS-CoV-2 severity in healthcare workers and patients | 24 months
  To investigate SARS-CoV-2 severity by review of any hospital admissions

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Ealing and Northwick Park hospital, London
  - The Francis Crick Institute, London
  - UCLH, London

REFERENCES:
- [Derived] Townsley H, Gahir J, Russell TW, Greenwood D, Carr EJ, Dyke M, Adams L, Miah M, Clayton B, Smith C, Miranda M, Mears HV, Bailey C, Black JRM, Fowler AS, Crawford M, Wilkinson K, Hutchinson M, Harvey R, O'Reilly N, Kelly G, Goldstone R, Beale R, Papineni P, Corrah T, Gilson R, Caidan S, Nicod J, Gamblin S, Kassiotis G, Libri V, Williams B, Gandhi S, Kucharski AJ, Swanton C, Bauer DLV, Wall EC. COVID-19 in non-hospitalised adults caused by either SARS-CoV-2 sub-variants Omicron BA.1, BA.2, BA.4/5 or Delta associates with similar illness duration, symptom severity and viral kinetics, irrespective of vaccination history. PLoS One. 2024 Mar 21;19(3):e0294897. doi: 10.1371/journal.pone.0294897. eCollection 2024. PMID 38512960